CLINICAL TRIAL: NCT06334900
Title: Retrospective Analysis of the French National Cohort of Patients With GAD Antibodies and Cerebellar Ataxia
Acronym: Ata-GAD
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0297
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: GAD-receptor Antibodies-associated Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-GAD encephalitis: This is a non-interventional study involving clinical data. This data are information of medical follow up on patient like diagnosis, symptoms, biological results, cancer, treatments.
  Interventions: Other: GAD patients

INTERVENTIONS:
Other: GAD patients — Describe the clinical and demographic characteristics of patients with anti-GAD65 antibody associated cerebellar ataxia.

SUMMARY:
Glutamic acid decarboxylase (GAD) is an enzyme whose function in the body is to decarboxylate glutamate to GABA. GAD65 antibodies (GAD65Ab) have been associated with type-1 diabetes (80% of new-onset patients) and various neurological conditions, mainly stiff-person syndrome (SPS/PERM), cerebellar ataxia (CA), limbic encephalitis (LE) and temporal lobe epilepsy. These syndromes all seem to result from a reduced transmission of GABA. These neurological conditions are rare and can cause symptoms like confusion, memory loss, muscle stiffness, muscle spasms, behavioural disorders, and pharmacoresistant epilepsy. When finding high levels of GAD65-Ab in the serum, a cerebrospinal fluid (CSF) sample should be taken to look for oligoclonal IgG bands and intrathecal GAD-Ab production to prove an auto-immune cause for the various neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* neurological symptoms with GAD antibody
* GAD antibody in sera and/or CSF
* patient with cerebellar ataxia

Exclusion Criteria:

* tested positive to another antibody.
* no data
* any test in paraneoplastic neurological syndrome and autoimmune encephalitis center

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with cerebellar ataxia and GAD antibody
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
GAD Patient | Baseline
  Description of clinical data in patients with cerebellar syndrome associated with anti-GAD antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique Pierre Wertheimer / Groupement Hospitalier Est, Bron, France